CLINICAL TRIAL: NCT02956213
Title: Assessing the Effect of Different Efficiency Indoor Air Filters on Respiratory Symptoms in Former Smokers
Brief Title: Indoor Air Quality and Respiratory Symptoms in Former Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1050302
Record Dates: First submitted 2016-10-19; First posted 2016-11-07 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; air filter; indoor air quality; respiratory symptoms; emphysema; chronic obstructive pulmonary disease; tobacco use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Signs and Symptoms, Respiratory; Emphysema; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM 1 MERV17 first (Experimental): This group will receive a portable HEPA air filtering device with MERV17 air filter for the first part of the study. At cross over, this group will receive the "placebo" or no high-efficiency filter.
  Interventions: Other: HEPA portable air filter
- ARM 2 MERV17 second (Active Comparator): This group will receive a HEPA portable air filter with no high efficiency air filter for the first part of the study. At cross over, this group will receive the high-efficiency MERV17 air filter.
  Interventions: Other: Sham Control/Active Comparator

INTERVENTIONS:
Other: HEPA portable air filter — A high efficiency (MERV17) portable air filter (HEPA portable air filter) will be placed in the subject's bedroom and will run 24/7 for the duration of the study.
  Arms: ARM 1 MERV17 first
Other: Sham Control/Active Comparator — A portable air filtering device will be placed with no high-efficiency air filter, but only the basic carbon filter in place. Then at cross over, there will be an active HEPA portable air filter used
  Arms: ARM 2 MERV17 second

SUMMARY:
The investigators will conduct a randomized, controlled, double-blind, crossover trial to determine whether the presence of a portable high-efficiency indoor air filter in the bedroom reduces respiratory symptoms in former smokers compared with placebo. The primary outcomes will be change in St. George's Respiratory Questionnaire - COPD (SGRQ-C) score associated with using a portable high-efficiency indoor air filter during the study period. Secondary outcomes of COPD exacerbations and hospitalizations, daily step counts, medication changes, spirometry, and cardiovascular outcomes will also be assessed.

DETAILED DESCRIPTION:
Hypothesis/Research Questions:

This study will determine whether the presence of a portable high-efficiency indoor air filter in the bedroom improves respiratory symptoms (based on St. George's Respiratory Questionnaire - COPD - SGRQ-C score) during a period of high air pollution compared with placebo in former smokers with respiratory symptoms.

The primary outcome will be the change in SGRQ-C score associated with using a portable high-efficiency indoor air filter during the study period.

Secondary outcomes will assess the effect of using a portable high-efficiency indoor air filter on healthcare utilization, other symptom scores, COPD exacerbation frequency, medication use, median daily step counts, inflammatory markers, oxygenation, indoor particulate counts and indoor-outdoor particulate count difference, and pulmonary function tests.

Baseline descriptive statistics will report baseline air filter type, duration of use, and particulate weight prior to study enrollment.

Evaluation of change in symptom scores and other secondary outcomes from baseline to study air filter (Visit 1 vs. Visit 2).

ELIGIBILITY:
Inclusion Criteria:

* history of smoking
* Do not currently smoke and no one currently smokes inside the home
* history of exacerbation or development of respiratory symptoms (e.g.cough, sputum production, chest tightness, exertional dyspnea, etc.) with periods of high outdoor air pollution ("inversions")
* Age 40 or older
* Access to Wi-Fi
* Access to a cell phone, tablet or personal computer

Exclusion Criteria:

* active tobacco use of subject
* active tobacco use in the home
* pre-existing use of a HEPA filter in the subject's bedroom

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-11; Primary Completion 2019-05-15 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in SGRQ-C score | 12 weeks
  based on St. George's Respiratory Questionnaire - COPD - SGRQ-C score

SECONDARY OUTCOMES:
Effect of air filtration on healthcare utilization | 6 months
  Effect on COPD related ER visits and hospitalizations; CHF and MI related visits and hospitalizations and all cause ER visits and hospitalizations
Aggregated assessment of the effect of air filtration on COPD exacerbation frequency | 6 months
  A combined assessment of patient reported symptom questionnaires including increased medication use, ER visits and hospitalizations for breathing-related problems and COPD exacerbations. These assessments will be determined by patient reported hospitalizations/ED visits, and patient reported symptom increase and COPD-related medication changes.
Change in median daily step counts | 6 months
  Whether median daily step counts are affected by air pollution levels, or correlate with other metrics of COPD outcomes remains unknown and thus, step counts will be tracked.
Change in inflammatory markers | 6 months
  This is a common office test used to assess how well the lungs work by measuring how much air the patients inhale, how much they exhale, and how quickly they exhale.
  We will also perform pulse oximetry and a blood draw to assess inflammatory markers and basic labs.
  COPD sufferers experience inflammation due to their disease. Inflammatory markers will be documented during their clinic visits.
Change in spirometry | 3 months
  Spirometry will be used to assess how well a subject's lungs work by measuring how much air is inhaled, how much is exhaled and how quickly you exhale. Spirometry is used to diagnose COPD and tracks it's progression or improve.
Number of cardiovascular events | 6 months
  CVA, MI, heart failure exacerbation
Change in 6 minute walk test | 3 months
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

OTHER OUTCOMES:
Change in sleep efficiency | 12 weeks
  As measured by the activity tracker, the amount of hours slept
Change in sleep quality | 12 weeks
  As measured by the activity tracker, the number of disruptions in sleep
Change in CAT scores | 12 weeks
  COPD assessment test is a questionnaire used to determine subjective improve or progression of COPD.
Change in mMRC scores | 12 weeks
  Modified Medical Research Council Dyspnea Scale score used to track a subject's shortness of breath
Change in other metrics of activity: specifically 6min walk distances and max walk distance | 12 weeks
  walk distance
Change in air filter changing habits | 12 months
  Change in air filter changing habits
Change in air filter weight with different filters (surrogate for particulates trapped) | 12 months
  Change in air filter weight with different filters (surrogate for particulates trapped)
Change in activity tracker use following study | 12 months
  Question in 6 month follow up from study if participants bought their own step counter or if they already had a step counter, if they use the device more as a result of the study.
Change in indoor particulate concentration as measured by personal air monitors (PurpleAir.org) | 3 months
  Change in indoor particulate concentration as measured by personal air

CONTACTS AND LOCATIONS:
Overall Officials: Denitza Blagev, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No